CLINICAL TRIAL: NCT07165626
Title: Evaluation of Morphological and Functional Changes in Eyes With Epiretinal Membrane After Vitrectomy
Brief Title: Evaluation of Retinal Parameters in Patients With Epiretinal Membrane After Vitrectomy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KB-006/25/2024
Record Dates: First submitted 2025-08-18; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Epiretinal Membrane; Macular Oedema; Macular Diseases; Retinal Diseases
MeSH Terms: conditions — Epiretinal Membrane; Macular Edema; Retinal Diseases

STUDY DESIGN:
Intervention Model Description: Parallel assignment with participants randomized 1:1 to either the laser-treated group or the control (nonlaser) group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser-treated group (Active Comparator): Additional subthreshold micropulse laser therapy (SMLT) using a 577 nm solid-state yellow diode laser, applied to the macular area (thirty 5 × 5 spot sizes of 160 µm, zero-spot spacing, including the fovea; fixed power 250 mW; exposure 200 ms; micropulse mode, 5% duty cycle) performed 1 month after pars plana vitrectomy (PPV).
  Interventions: Device: Subtreshold micropulse laser therapy; Procedure: Pars plana vitrectomy
- Nonlaser group (Other): Pars plana vitrectomy (PPV) performed without subsequent subthreshold micropulse laser therapy (SMLT).
  Interventions: Procedure: Pars plana vitrectomy

INTERVENTIONS:
Device: Subtreshold micropulse laser therapy — Laser-treated group will receive additional subthreshold micropulse laser therapy (SMLT) 1 month after pars plana vitrectomy (PPV), using a 577 nm solid-state yellow diode laser applied to the macular area (thirty 5 × 5 spot sizes of 160 µm, zero-spot spacing, including the fovea; fixed power 250 mW; exposure time 200 ms; micropulse mode, 5% duty cycle). Control group (nonlaser group) will not receive additional laser treatment.
  Arms: Laser-treated group
Procedure: Pars plana vitrectomy — Both groups will undergo pars plana vitrectomy (PPV) with epiretinal membrane (ERM) and internal limiting membrane (ILM) peeling prior to allocation to study arms.

SUMMARY:
The goal of this interventional study is to assess the dynamics of structural and functional retinal changes in eyes with epiretinal membrane (ERM) after pars plana vitrectomy (PPV). Other study objectives include:

* Identification of preoperative prognostic factors associated with better postoperative outcomes.
* Evaluation of the utility of advanced, highly specialized retinal function testing as diagnostic-prognostic tools in patients after ERM surgery.
* Definition of updated qualification criteria and surgical indications for vitrectomy in patients with ERM.

Researchers will compare a laser-treated group (additional subthreshold micropulse yellow laser (577 nm) at 1 month post-PPV) with a nonlaser group (no additional laser) to see whether early postoperative subtreshold micropulse laser therapy (SMLT) affects selected functional and morphometric retinal parameters after ERM peeling.

This prospective, randomized, controlled, single-center study includes 100 pseudophakic patients scheduled for surgical ERM removal.

Eligibility requires a visually significant ERM with metamorphopsia and/or reduced best-corrected visual acuity.

Participants are classified preoperatively by OCT-based Govetto staging and randomized 1:1 to either the laser-treated group or the non-laser (control) group. All patients undergo standard 25-gauge PPV with ERM peeling, followed by ILM peeling and SF₆ gas tamponade, performed by a single experienced vitreoretinal surgeon.

Follow-up visits occur preoperatively, and at 1 and 4 months postoperatively; SMLT is performed at 1 month in the laser arm. Baseline questionnaire captures metamorphopsia presence (yes/no) and duration (<6, 6-12, >12 months).

Assessments include:

* best corrected visual acuity (BCVA) [Snellen and ETDRS charts]
* enhanced depth imaging optical coherence tomography (EDI-OCT) [retinal thickness in the nine Early Treatment Diabetic Retinopathy Study (ETDRS) subfields (μm); total retinal volume (mm³); subfoveal choroidal thickness (μm); choroidal area (mm²)]
* OCT angiography (OCTA) [foveal avascular zone (FAZ) area in both the superficial (SVC) and deep vascular complexes (DVC) (mm²)]
* multifocal electroretinography (mfERG) [P1-wave retinal response density (nV/deg²) in rings R1-R6; P1-wave implicit (peak) time in rings R1-R6 (ms)]
* microperimetry (average threshold (dB); fixation stability P1/P2; fixation variability via 63% and 95% bivariate contour ellipse area (BCEA)]
* wide-field fundus imaging

Statistical analyses will be performed at a significance level of p<0.05, using appropriate parametric or nonparametric methods selected based on data distribution and measurement scale.

ELIGIBILITY:
Inclusion Criteria:

* Epiretinal membrane (ERM) - either associated with metamorphopsia or causing a marked reduction in best corrected visual acuity
* Pseudophakia

Exclusion Criteria:

* Coexisting ocular or retinal diseases other than ERM
* Evidence of ocular inflammation or any active intraocular inflammatory process

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in BCVA from 1 month post-PPV (pre-laser) to 4 months post-PPV. | 1 month (pre-laser) and 4 months postoperatively.
  Between-group difference (laser-treated group vs nonlaser group) in change in best corrected visual acuity (BCVA) from Month 1 to Month 4. BCVA measured using Snellen and ETDRS charts.

SECONDARY OUTCOMES:
Change in mfERG P1-wave retinal response density in rings R1-R6. | Baseline (pre-op), 1 month, and 4 months post-op.
  Multifocal electroretinography (mfERG) P1-wave retinal response density (nV/deg²) in rings R1-R6. Analyses will include between-group changes from Month 1 to Month 4 and overall within-subject changes from baseline to Month 1 and from baseline to Month 4 (across both arms).
Change in mfERG P1-wave implicit time in rings R1-R6. | Baseline (pre-op), 1 month, and 4 months post-op.
  Multifocal electroretinography (mfERG) P1-wave implicit (peak) time (ms) in rings R1-R6. Analyses will include between-group changes from Month 1 to Month 4 and overall within-subject changes from baseline to Month 1 and from baseline to Month 4 (across both arms).
Change in average threshold on microperymetry. | Baseline (pre-op), 1 month, and 4 months post-op.
  Average threshold (dB) on microperymetry. Analyses will include between-group changes from Month 1 to Month 4 and overall within-subject changes from baseline to Month 1 and from baseline to Month 4 (across both arms).
Change in fixation stability P1 and P2 on microperymetry. | Baseline (pre-op), 1 month, and 4 months post-op.
  Fixation stability P1 and P2 (%) on microperymetry. Analyses will include between-group changes from Month 1 to Month 4 and overall within-subject changes from baseline to Month 1 and from baseline to Month 4 (across both arms).
Change in fixation variability on microperymetry. | Baseline (pre-op), 1 month, and 4 months post-op.
  Fixation variability via 63% and 95% bivariate contour ellipse area (BCEA) on microperymetry (deg²). Analyses will include between-group changes from Month 1 to Month 4 and overall within-subject changes from baseline to Month 1 and from baseline to Month 4 (across both arms).
Change in retinal thickness on EDI-OCT. | Baseline (pre-op), 1 month, and 4 months post-op.
  Retinal thickness in the nine Early Treatment Diabetic Retinopathy Study (ETDRS) subfields (μm) on enhanced depth imaging optical coherence tomography (EDI-OCT). Analyses will include between-group changes from Month 1 to Month 4 and overall within-subject changes from baseline to Month 1 and from baseline to Month 4 (across both arms).
Change in total retinal volume on EDI-OCT. | Baseline (pre-op), 1 month, and 4 months post-op.
  Total retinal volume (mm³) on EDI-OCT. Analyses will include between-group changes from Month 1 to Month 4 and overall within-subject changes from baseline to Month 1 and from baseline to Month 4 (across both arms).
Change in subfoveal choroidal thickness on EDI-OCT. | Baseline (pre-op), 1 month, and 4 months post-op.
  Subfoveal choroidal thickness (μm) on EDI-OCT. Analyses will include between-group changes from Month 1 to Month 4 and overall within-subject changes from baseline to Month 1 and from baseline to Month 4 (across both arms).
Change in choroidal area on EDI-OCT. | Baseline (pre-op), 1 month, and 4 months post-op.
  Choroidal area (mm²) on EDI-OCT. Analyses will include between-group changes from Month 1 to Month 4 and overall within-subject changes from baseline to Month 1 and from baseline to Month 4 (across both arms).
Change in FAZ area in the SVC and DVC on OCTA. | Baseline (pre-op), 1 month, and 4 months post-op.
  Foveal avascular zone (FAZ) area in the superficial vascular complex (SVC) (mm²) and deep vascular complex (DVC) (mm²) on OCT angiography (OCTA). Analyses will include between-group changes from Month 1 to Month 4 and overall within-subject changes from baseline to Month 1 and from baseline to Month 4 (across both arms).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Machalińska, Prof., MD, PhD, Principal Investigator — First Department of Ophthalmology, Pomeranian Medical University in Szczecin, Poland
Locations (1):
- First Department of Ophthalmology, Pomeranian Medical University, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: No